CLINICAL TRIAL: NCT03571321
Title: Phase I Trial of Ruxolitinib in Combination With a Pediatric Based-regimen for Adolescents and Young Adults (AYAs) With Ph-like Acute Lymphoblastic Leukemia (ALL)
Brief Title: Ruxolitinib and Chemotherapy in Adolescents and Young Adults With Ph-like Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-1110
Record Dates: First submitted 2018-06-22; First posted 2018-06-27 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphoblastic Leukemia; ALL, Childhood; ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ruxolitinib; Cyclophosphamide; Cytarabine; Mercaptopurine; Vincristine; pegaspargase; Rituximab; Methotrexate; Administration, Intravenous; Dexamethasone; Doxorubicin; Thioguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): Participants will receive ruxolitinib in addition to standard chemotherapy.
  Standard Chemotherapy Consists of:
  * Remission consolidation therapy (lasting 8 weeks)
  * Interim Maintenance (lasting 8 weeks)
  * Delayed Intensification (lasting 8 weeks
  * Maintenance Therapy (12 week courses/84 day cycles lasting 2-3 years)
  Prior to study entry, patients must have completed a 4-drug induction therapy regimen with intrathecal chemotherapy (modified Berlin-Frankfurt-Münster (aBFM) regimen or equivalent) as per the institution standard of care.
  Interventions: Drug: Ruxolitinib; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Vincristine; Drug: Pegaspargase; Drug: Rituximab; Drug: Methotrexate (Intrathecal Administration); Drug: Methotrexate (Intravenous Administration); Drug: Dexamethasone; Drug: Doxorubicin; Drug: Thioguanine; Drug: Methotrexate Oral Product

INTERVENTIONS:
Drug: Ruxolitinib — Participants will receive one of 3 doses [taken by mouth] (30 mg, 40 mg, or 50 mg) depending on when they are enrolled to the study.
  Remission consolidation regimen:
  * Days 1-14 and 29-43
  Interim maintenance regimen:
  * Days 1-14 and 29-43
  Delayed Intensification regimen:
  * Days 1-14 and 29-43
  Other Names: Jakafi
Drug: Cyclophosphamide — Remission consolidation regimen:
  * 1000 mg/m2 by intravenous infusion (IV) on Day 1 and Day 29
  Delayed Intensification regimen:
  * 1000 mg/m2 IV on Day 29
Drug: Cytarabine — Remission consolidation regimen:
  * 75 mg/m2/day IV or subcutaneously (SC) on Days 1-4 (i.e., 4 doses), 8-11, 29-32, and 36-39
  Delayed Intensification regimen:
  * 75 mg/m2/day IV or SC on Days 29-32 and 36-39
Drug: Mercaptopurine — Taken by mouth.
  Remission consolidation regimen:
  * 60 mg/m2 on Days 1-14 and 29-42
  Maintenance Therapy:
  * 75 mg/m2 on Days 1-84
Drug: Vincristine — Remission consolidation regimen:
  * 1.5 mg/m2 (maximum 2 mg) IV once per week on Days 15, 22, 43, and 50
  Interim maintenance regimen:
  * 1.5 mg/m2 (maximum 2 mg) IV on Days 1, 11, 21, 31, and 41
  Delayed Intensification regimen:
  * 1.5 mg/m2 (maximum 2 mg) IV on Days 1, 8, 15, 43, and 50
  Maintenance Therapy:
  * 1.5 mg/m2 (maximum 2 mg) IV on Days 1, 29, and 57
Drug: Pegaspargase — Remission consolidation regimen:
  * 2500 IU/m2 given by intramuscular (IM) injection or IV on Days 15 and 43
  Interim maintenance regimen:
  * 2500 IU/m2 IM or IV on Days 2 and 22
  Delayed Intensification regimen:
  * 2500 IU/m2 IM or IV on Day 4 (OR Day 5 OR Day 6) AND Day 43.
Drug: Rituximab — For patients that have cluster of differentiation antigen 20 positive (CD20+) disease only.
  Remission consolidation regimen:
  * 375 mg/m2 IV on Days 1, 8, 29 and 36
  Interim maintenance regimen:
  * 375 mg/m2 IV on Days 1 and 11
  Delayed Intensification regimen:
  * 375 mg/m2 IV on Days 1 and 8
Drug: Methotrexate (Intrathecal Administration) — Drug is given through a needle which is inserted in one of the spaces between the bones in the lower back (intrathecal [IT] administration).
  Remission consolidation regimen:
  * 15 mg on Days 1, 8, 15, and 22
  Interim maintenance regimen:
  * 15 mg on Days 1 and 31
  Delayed Intensification regimen:
  * 15 mg on Days 1, 29, and 36
  Maintenance Therapy:
  * 15 mg on Day 1
  * 15 mg on Day 29 (First 4 courses only)
Drug: Methotrexate (Intravenous Administration) — Interim maintenance regimen:
  * 100 mg/m2 IV on Days 1, 11, 21, 31, and 41
Drug: Dexamethasone — Taken by mouth or given by IV infusion.
  Delayed Intensification regimen:
  * 10 mg/m2 per day (divided into 2 doses) on Days 1-7 and 15-21
  Maintenance Therapy:
  * 6 mg/m2 per day (divided into 2 doses) on Days 1-5, 29-33, and 57-61
Drug: Doxorubicin — Delayed Intensification regimen:
  * 25 mg/m2 IV on Days 1, 8, 15
Drug: Thioguanine — Taken by mouth at least 1 hour after evening meal.
  Delayed Intensification regimen:
  * 60 mg/m2 on Days 29-42
Drug: Methotrexate Oral Product — Taken by mouth.
  Maintenance Therapy:
  * 20 mg/m2 weekly (on Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78)
  * Not given on Day 29 of first 4 courses (on days when IT Methotrexate is given]

SUMMARY:
This study will test if adding ruxolitinib to standard multi-drug chemotherapy regimen will be safe and tolerated in adolescents and young adults with newly diagnosed Ph-like acute lymphoblastic leukemia (ALL).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed de novo B-precursor acute lymphoblastic leukemia (ALL) as determined by World Health Organization (WHO) criteria. Patients must have unequivocal diagnosis of precursor B ALL. This includes an institutional immunophenotyping report that is to assign B-lineage or T-lineage.
* "Ph-like" signature, as determined by low density micro-array (LDA) card
* Jak-targetable genetic signature as defined by any of the following:

  * Cytokine receptor-like factor 2 (CRLF2) rearranged (JAK2 mutant or wild-type)
  * JAK2 or erythropoietin receptor (EPOR) fusions.
  * Other JAK pathway alterations at the discretion of the principle investigator including, but not limited to:
* SH2B adaptor protein 3 (SH2B3) deletions
* Interleukin-7 receptor subunit alpha (IL7RA) mutations
* Prior therapy

  * Prior to starting ruxolitinib, patients must have completed a 4-drug induction regimen with intrathecal chemotherapy (modified aBFM regimen or equivalent) as per the institutional standard of care. Recommended induction treatment is outlined in Section 5.1.2.
  * No additional prior therapy for acute leukemia except emergency therapy (corticosteroids or hydroxyurea) for blast cell crisis, superior vena cava syndrome, or renal failure due to leukemic infiltration of the kidneys. When indicated, leukapheresis or exchange transfusion is recommended to reduce the white blood cell count (WBC).
  * Screening may occur at any point prior to or during induction therapy
* Age ≥ 18 years and < 40 years. Because this is specifically a study of the adolescent and young adult population and no adverse event data are currently available on the use of this pediatric-based chemotherapy regimen in patients ≥ 40 years of age, older adults are excluded from this study, but may be eligible for future trials.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥ 60%)
* Platelet count > 25,000/uL.
* Patients must have normal organ function as defined below:

  * total bilirubin ≤ 2 mg/dL
  * aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ≤ 2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Because the therapeutic agents used in this study are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who are receiving any other investigational agent.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 3 years.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ruxolitinib or other agents used in study.
* Use of any potent cytochrome P450 (CYP) 3A4 inhibitor or inducer within 5 half-lives before the first dose of the study drug. Potent inhibitors of CYP3A4 include systemic ketoconazole, posaconazole, voriconazole, clarithromycin, itraconazole, nefazodone, and telithromycin. At the fluconazole dose of 200mg daily used this regimen, there is minimal inhibition of CYP3A4 [36] and therefore fluconazole is not prohibited on this trial and no dose modifications should be made in the presence of fluconazole.

Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because ruxolitinib is a class C agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ruxolitinib breastfeeding should be discontinued if the mother is treated with ruxolitinib. These potential risks may also apply to other agents used in this study.
* Down Syndrome due to the likelihood of excessive toxicity resulting. These patients should be treated in consultation with a pediatric oncologist.
* Burkitt type leukemia
* Ph+ ALL at time of diagnosis

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of adding ruxolitinib to a standard-of-care pediatric-based chemotherapy regimen in adolescents and young adult patients as determined by rate of side effects seen when combination is given | 24 weeks
  Determined by rate of side effects seen when combination is given

SECONDARY OUTCOMES:
Rate of participants that are minimal residual disease (MRD) negative at end of induction therapy | 4 weeks
Overall survival rate | 2 years
Event-free survival rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Stock, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States